CLINICAL TRIAL: NCT06494644
Title: An Open-label, Single-group, Three-period, Fixed-sequence, Phase I Study to Assess the Pharmacokinetics of AZD6793 Tablets When Administered Alone and in Combination With Itraconazole Capsules in Healthy Adult Female and Male Participants.
Brief Title: A Study to Assess the Pharmacokinetics of AZD6793 When Administered Alone and in Combination With Itraconazole in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D7860C00004; 2023-509002-30-00 (Other: EU-CT number)
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
Keywords: AZD6793; Itraconazole; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-group, 3 period fixed sequence study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD6793 and Itraconazole (Experimental): Participants will receive a single dose of AZD6793 on Day 1. On Day 4, the participant will receive 2 doses of 200 mg itraconazole 12 hours apart followed by a single dose of 200 mg itraconazole from Days 5 to 7. On Day 8, participants will receive a combined dose of AZD6793 and 200 mg itraconazole. On Day 9 and Day 10, the participants will receive a single dose of 200 mg itraconazole.
  Interventions: Drug: AZD6793; Drug: Itraconazole; Drug: AZD6793+ Itraconazole

INTERVENTIONS:
Drug: AZD6793 — Participants will receive single dose of AZD6793 on Day 1 in Period 1 and on Day 8 in combination with itraconazole in Period 3.
Drug: Itraconazole — Participants will receive 2 doses of itraconazole on Day 4 and single dose from Day 5 to Day 7 in Period 2. On Day 8 participants will receive single dose of itraconazole combined with AZD6793 and then single dose of itraconazole from Day 9 to Day 10 in Period 3.
Drug: AZD6793+ Itraconazole — Participants will receive a combined dose of AZD6793 and itraconazole on Day 8 in Period 3.

SUMMARY:
The study will evaluate the pharmacokinetics (PK) of AZD6793 when administered alone and in combination with itraconazole in healthy adult participants.

DETAILED DESCRIPTION:
This is a single-group study with a duration of up to 8 weeks (maximum of 53 days) including Screening, Period 1, Period 2, Period 3 and Follow-up.

The study will comprise of:

* A screening period of 27 days
* Three treatment periods: Period 1 (Day -1 to Day 3): Single dose AZD6793 will be administered on Day 1 followed by a 3-day washout period; Period 2 (Day 4 to Day 7): Itraconazole will be administered from Day 4 through Day 7, starting with 2 doses of 200 mg itraconazole given 12 hours apart on Day 4, then 200 mg itraconazole will be given once a day on Day 5 through Day 7. Period 3 (Day 8 to Day 11): On Day 8, participants will be co-administered with AZD6793 and 200 mg itraconazole. Administration of 200 mg itraconazole will continue on Day 9 and Day 10. Participants will be discharged from the clinic on Day 11.
* A Follow-up Visit 10-15 days after the last itraconazole dose in Period 3.

ELIGIBILITY:
Main Inclusion Criteria:

* Female participants must have a negative pregnancy test at screening and on admission and must not be lactating.
* Females of childbearing potential must not be lactating and, if heterosexually active, must agree to use with their partner an approved method of highly effective contraception to avoid pregnancy.
* Females of non-childing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods from Screening visit until 3 months after Follow-up visit.
* Participants with Body mass index between 18 and 30 kg/m², and at least 50 kg at the Screening Visit.
* Participants should be fully/sufficiently vaccinated against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) as per current local regulations.

Main Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, renal, or pancreatic disease, or any other clinically significant disease or disorder known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of clinically significant chronic or active hematologic disease.
* Diagnosis or history of immunodeficiency or increased susceptibility to severe infection, or a clinically significant infection within 4 weeks of the Screening Visit.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug.
* Any laboratory values with deviations at the Screening Visit or on admission to the Clinical Unit. Abnormal values may be repeated at the discretion of the Investigator: Alanine transaminase (ALT) > Upper Limit Normal (ULN), Aspartate Transaminase (AST) > ULN, WBC count < Lower limit normal (LLN), Neutrophils > ULN or < LLN, Haemoglobin < 120 g/L, Bilirubin > ULN, Urinary albumin to creatinine ratio abnormal (≥ 3.4 mg/mmol), eGlomerular filtration rate (eGFR) < 85 mL/min/1.73 m² calculated using the CKD-EPI equation (eGFR will only be assessed at Screening).
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results at the screening.
* Positive or indeterminate QuantiFERON® TB test at the Screening Visit.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, or Human immunodeficiency virus (HIV).
* Participants with a history or presence of vitiligo or significant (in the opinion of the investigator) skin depigmentation for any cause including drugs.
* Any clinically significant abnormal finding in vital signs, at the Screening Visit and/or on admission to the Clinical Unit.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse, alcohol, or cotinine (nicotine) at screening visit or on admission to the Clinical Unit.
* History or presence of severe allergy/hypersensitivity.
* Excessive intake of caffeine-containing drinks or food.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of the study drug.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of >3 times the recommended daily dose) and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of study drug. The use of hormonal replacement therapy for females is not permitted.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of study intervention in this study.
* Participants who have previously received AZD6793.
* Vulnerable participants.
* Participant has a positive test result for SARS-CoV-2 via RT-PCR on admission to the Clinical Unit.
* Participant has clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19).
* Participant who had severe course of COVID-19.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Maximum plasma drug concentration (Cmax) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose Cmax of AZD6793 will be evaluated in healthy participants.
Area under plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose AUClast of AZD6793 will be evaluated in healthy participants.
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose AUCinf of AZD6793 will be evaluated in healthy participants.
Apparent total body clearance (CL/F) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose CL/F of AZD6793 will be evaluated in healthy participants.
Terminal elimination half-life (t1/2λz) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose t1/2λz of AZD6793 will be evaluated in healthy participants.
Time to reach maximum observed concentration (tmax) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose tmax of AZD6793 will be evaluated in healthy participants.
Apparent volume of distribution during the terminal phase (Vz/F) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose Vz/F of AZD6793 will be evaluated in healthy participants.
Ratio Area under plasma concentration-time curve from time 0 to infinity (RAUCinf) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose RAUCinf of AZD6793 will be evaluated in healthy participants.
Ratio Area under plasma concentration-time curve from time 0 to the last quantifiable concentration (RAUClast) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose RAUClast of AZD6793 will be evaluated in healthy participants.
Ratio Maximum plasma drug concentration (RCmax) | Post-dose on Day 1 to Day 3; and Day 8 to Day 11
  The effect of itraconazole on the single-dose RCmax of AZD6793 will be evaluated in healthy participants.

SECONDARY OUTCOMES:
Number of participants with adverse events | From first dose (Day 1) until Follow-up (10-15 days post last itraconazole dose)
  The safety and tolerability after administration of AZD6793 with itraconazole will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/